CLINICAL TRIAL: NCT02702622
Title: Vitamin A Equivalence of the Provitamin A in Biofortified Bananas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Wendy S. White, Associate Professor, Iowa State University
Other Study IDs: 13-376
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Vitamin A Deficiency
Keywords: bananas; biofortified; carotenoids; vitamin A
MeSH Terms: conditions — Vitamin A Deficiency

INTERVENTIONS:
Other: Provitamin A-biofortified transgenic bananas

SUMMARY:
The objective will be to quantify the vitamin A equivalence of the provitamin A in transgenic biofortified bananas.

ELIGIBILITY:
Inclusion Criteria:

* General good health as determined by interview, blood biochemistry profile, and complete blood count
* Antecubital veins amenable to blood collection

Exclusion Criteria:

* Adverse reactions to blood sample collection
* History of anemia or excessive bleeding
* Cigarette smoking, frequent alcohol consumption
* Use of vitamin/mineral supplements
* Food allergies
* Lactose intolerance
* Abnormal thyroid status
* Chronic disease, lipid malabsorption or gastrointestinal disorders
* Hyper- or hypolipidemia
* Body mass index (BMI) > 28
* History of eating disorder or restrained eating
* Current or planned pregnancy; menstrual cycle irregularities or abnormalities
* Use of hormonal contraceptives (affects chylomicron clearance); use of medications that may affect lipid absorption or transport

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2016-03; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve for retinyl ester in the plasma triacylglycerol-rich lipoprotein fraction | 0 - 9.5 hours postprandially